CLINICAL TRIAL: NCT07378241
Title: Observation of the Effect of Patients' Hormone Levels on Sedoanalgesia in Oocyte Pcik-Up: Prospective Observational Study
Brief Title: Effects of Patients' Hormone Levels on Sedoanalgesia
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Gözde Gürsoy Çirkinoğlu, MD, Izmir City Hospital
Other Study IDs: Oocyte Pick Up
Record Dates: First submitted 2025-05-26; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Consumption of Anaesthetic Agents; Sedoanalgesia
Keywords: sedoanalgesia; OPU; Progesterone; estrogen

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OPU patients: patients progesteron estrogen levels and progesteron/estrogen ratios
  Interventions: Drug: Anesthesia Maintenance

INTERVENTIONS:
Drug: Anesthesia Maintenance — the amount of propofol required to achieve depth of anaesthesia in mg/kg/minute

SUMMARY:
Investigastors hypothesis is that the need for anaesthetic agents is less in patients with high progesterone levels and more in patients with high estrogen levels.

DETAILED DESCRIPTION:
In anaesthesia practice, the need for anaesthetic agents can be affected by many different factors. These factors may include age, gender, body weight, existing hepatic or renal insufficiency, cardiovascular diseases, low ejection fraction, and some hormonal changes may also be effective in the need for anaesthetic agents. For example, there are studies showing that progesterone, which increases in the last period of pregnancy in pregnant women, decreases the use of anaesthetic agents due to its central effects. In a study by, the MAC level of sevoflurane was measured by following the haemodynamic data and bispectral indexes of the patients and the amount of sevoflurane used was found to be less in patients with higher serum progesterone levels in pregnant women with gestational pregnancies older than 36 weeks undergoing planned cesarean section.

Estrogen and progesterone ratios regulate gonadotropin secretion and sexual behaviour in the brain. In addition, although it is known to be effective in analgesia and pain sensation pathways, this mechanism has not yet been fully understood . In an experimental animal study, it was concluded that estrogen facilitates pain transmission in acute pain pathways. In an animal study conducted in female rats, the need for anaesthetic agent in anaesthesia practice can be affected by many different factors at different times of the menstrual cycle phases. These factors may include age, gender, body weight, existing hepatic or renal insufficiency, cardiovascular diseases, low ejection fraction, and some hormonal changes may also be effective in the need for anaesthetic agents. For example, there are studies showing that progesterone, which increases in the last period of pregnancy in pregnant women, decreases the use of anaesthetic agents due to its central effects. In a study, the MAC level of sevoflurane was measured by following the haemodynamic data and bispectral indexes of the patients and the amount of sevoflurane used was found to be less in patients with higher serum progesterone levels in pregnant women with gestational pregnancies older than 36 weeks undergoing planned cesarean section.

Estrogen and progesterone ratios regulate gonadotropin secretion and sexual behaviour in the brain. In addition, although it is known to be effective in analgesia and pain sensation pathways, this mechanism has not yet been fully understood. In an experimental animal study, it was concluded that estrogen facilitates pain transmission in acute pain pathways. In an animal study in female rats, it was concluded that the characteristics of mu receptors in the brain changed in relation with the amounts of estrogen and progesterone secretion at different times of menstrual cycle phases. There are many publications in the literature examining the effects of estrogen and progesterone on analgesia pathways.

In today's anaesthesia practice, we encounter a large number of female patients both in operation theatres and in daily anaesthesia. In the process of in vitro fertilisation treatments, which is one of these areas, the need for daily anaesthesia arises for many procedures. Especially oocyte collection is performed with sedational procedures. Before the oocyte collection procedure, various hormone supplements are administered to the patients to ensure oocyte maturation, and patients who are shown to have reached adequate hormone levels in the laboratory with pre-procedure USG examination are taken to the oocyte collection procedure for aspiration of the follicles formed. This procedure requires a level of sedation in which patients can be immobilised and painless.

Investigastors hypothesis is that the need for anaesthetic agents is less in patients with high progesterone levels and more in patients with high estrogen levels.

The investigators' plan in this study is to examine the correlations of progesterone level, estrogen level, progesterone/estrogen level parameters with anaesthetic agent consumption via 3 groups

ELIGIBILITY:
Inclusion Criteria:

* Between 18-45 years old
* ASA-I ASA-II patients who were sedated for oocyte pick-up between 1 June 2025 and 1 September 2025 at Izmir City Hospital
* Patients whose hormone levels were measured in the preoperative period due to surgical indication and registered in the hospital data processing system

Exclusion Criteria:

* Lack of patient approvel
* Diagnosed psychiatric disorder
* Use of drugs affecting the central nervous system
* Presence of chronic pain syndrome
* History of continuous analgesic use due to chronic pain
* Hepatic and/or renal insufficiency
* BMI>30
* Changing the method of anaesthesia for any reason

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Between 18-45 years old
  * ASA-I ASA-II patients who were sedated for oocyte pick-up between 1 June 2025 and 1 September 2025 at Izmir City Hospital
  * Patients whose hormone levels were measured in the preoperative period due to surgical indication and registered in the hospital data processing system
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Anesthetic consumptiom | intraoperative
  the amount of propofol needed to provide adequate depth of anaesthesia in mg/kg/minute

SECONDARY OUTCOMES:
Pulse oximeter | intraoperative
  pulse oksimeter values at the begining, 10 minutes later and final
hearth rate changes | intraoperative
  Heart rate (bp/min) at the begining, 10 minutes later, final
Blood pressure changes | intraoperative
  Blood pressure values (mm/Hg) at the begining, 10 minutes later, final

CONTACTS AND LOCATIONS:
Overall Officials: Halide Hande Şahinkaya, MD, Study Chair — Izmir City Hospital, Anesthesiology and Reanimation Department; Tuba Kuvvet Yoldaş, MD, Study Chair — Izmir City Hospital, Anesthesiology and Reanimation Department; Zeki Tuncer Tekgul, Prof. Dr., Study Chair — Izmir City Hospital, Anesthesiology and Reanimation Department

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee J, Lee J, Ko S. The relationship between serum progesterone concentration and anesthetic and analgesic requirements: a prospective observational study of parturients undergoing cesarean delivery. Anesth Analg. 2014 Oct;119(4):901-905. doi: 10.1213/ANE.0000000000000366. PMID 25036373